CLINICAL TRIAL: NCT00006215
Title: A Phase II Study of Docetaxel and Vinorelbine in Advanced Non-Small Cell Lung Carcinoma
Brief Title: Docetaxel and Vinorelbine Plus Filgrastim in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amgen (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067941; AMGEN-GCSF-990138; NCI-V00-1596
Record Dates: First submitted 2000-09-11; First posted 2004-03-17 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-12

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Filgrastim; Docetaxel; Vinorelbine

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus filgrastim in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response to docetaxel and vinorelbine with filgrastim (G-CSF) support in patients with stage IIIB or IV non-small cell lung cancer. II. Determine the toxicity of this regimen in these patients. III. Determine the overall survival and time to tumor progression in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive vinorelbine IV over 6-10 minutes and docetaxel IV over 1 hour on day 1 and filgrastim (G-CSF) subcutaneously daily on days 2-12 or until blood counts recover. Treatment continues every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer Bidimensionally measurable or evaluable disease No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 70-100% Life expectancy: Greater than 2 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: AST and ALT no greater than 1.5 times upper limit of normal (ULN) Bilirubin no greater than ULN Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No uncontrolled hypertension, unstable angina, congestive heart failure, or atrial or ventricular arrhythmias At least 6 months since prior myocardial infarction Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No poorly controlled diabetes No known allergy to E. coli derivatives or any products to be administered No other prior malignancy within the past 5 years except surgically cured basal cell skin cancer or carcinoma in situ of the cervix No active infection or fever Not previously entered in this study

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent hematopoietic growth factors Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy and recovered Surgery: At least 2 weeks since prior major thoracic or abdominal surgery and recovered At least 6 months since prior coronary angioplasty Other: At least 30 days since prior investigational agents No other concurrent investigational agent No prophylactic acetaminophen for fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Allen, DVM, MBA, PharmD, Study Chair — Amgen
Locations (19):
- United States (19):
  - Gould Medical Group, Modesto, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Georgia Cancer Treatment Center, P.C., Riverdale, Georgia
  - Oncology and Hematology Associates, Westwood, Kansas
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Hematology-Oncology Associates of Rockland, P.C., New City, New York
  - New York Medical College, Valhalla, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group, Independence, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Trident Palmetto Hematology/Oncology, North Charleston, South Carolina
  - Boston Baskin Cancer Group, University Tennessee Oncology/Hematology Group, Memphis, Tennessee
  - Texas Cancer Care, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Hematology & Oncology Associates of Virginia, Richmond, Virginia
  - Morgantown Internal Medicine Group, Morgantown, West Virginia